CLINICAL TRIAL: NCT02412982
Title: Evaluation of Venous Thromboembolism Prevention in High-Risk Trauma Patients: A Prospective Randomized Trial of Standard Enoxaparin Versus Two Anti-Xa Adjusted Dosing Strategies
Brief Title: Evaluation of Venous Thromboembolism Prevention in High-Risk Trauma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Molly Droege, Clinical Pharmacy Specialist, Trauma, Surgery, and Orthopedics, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Droege2015
Record Dates: First submitted 2015-02-24; First posted 2015-04-09 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Traumatic Injury; Venous Thromboembolism
MeSH Terms: conditions — Wounds and Injuries; Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Serum anti-Xa >= 0.1 IU/mL (No Intervention): Patients with serum anti-Xa level >= 0.1 IU/mL after third dose of enoxaparin 30 mg every 12 hours
- Anti-Xa <0.1 IU/mL:enoxaparin 40 mg q12h (Active Comparator): Patients with serum anti-Xa level < 0.1 IU/mL after third dose of enoxaparin 30 mg every 12 hours who then receive enoxaparin 40 mg every 12 hours. If repeat steady state trough anti-Xa is subtherapeutic, dose will be increased to enoxaparin 50 mg every 12 hours.
  Interventions: Drug: Enoxaparin 40 mg q12h
- Anti-Xa <0.1 IU/mL:enoxaparin 30 mg q8h (Active Comparator): Patients with serum anti-Xa level < 0.1 IU/mL after third dose of enoxaparin 30 mg every 12 hours who then receive enoxaparin 30 mg every eight hours
  Interventions: Drug: Enoxaparin 30 mg q8h
- Serum anti-Xa < 0.1 IU/mL (No Intervention): Patients with serum anti-Xa level < 0.1 IU/mL after third dose of enoxaparin 30 mg every 12 hours

INTERVENTIONS:
Drug: Enoxaparin 40 mg q12h — Patients receive enoxaparin 40 mg every 12 hours. Dose will be escalated to enoxaparin 50 mg every 12 hours if steady state trough concentration is still subtherapeutic.
  Other Names: no other name
  Arms: Anti-Xa <0.1 IU/mL:enoxaparin 40 mg q12h
Drug: Enoxaparin 30 mg q8h — Patients receive enoxaparin 30 mg every 8 hours.
  Other Names: no other name
  Arms: Anti-Xa <0.1 IU/mL:enoxaparin 30 mg q8h

SUMMARY:
This is a pilot study to determine if anti-thrombin III (AT-III) serum concentrations differ between patients with normal versus subtherapeutic anti-Xa trough concentrations when placed on enoxaparin 30 mg twice daily for VTE prophylaxis. Secondarily, this study will compare two enoxaparin dosing strategies.

DETAILED DESCRIPTION:
This is a pilot study to determine if AT-III serum concentrations differ between patients with normal (>= 0.1 IU/mL) versus subtherapeutic (<0.1 IU/mL) anti-Xa trough concentrations when placed on enoxaparin 30 mg twice daily for venous thromboembolism (VTE) prophylaxis. Secondarily, this study will compare two enoxaparin dosing strategies: standard 30 mg twice daily and a dosing strategy based on trough anti-Xa values in high-risk trauma patients.

Specific aims include: 1) to compare the extent of reduced AT-III activity between patients with trough anti-Xa >= 0.1 IU/mL and < 0.1 IU/mL upon initial assay; 2) to determine the proportion of patients who reach goal anti-Xa and the time to goal anti-Xa achievement between two interventional dosing strategies: enoxaparin 40 mg every 12 hours (with consideration to increase to 50 mg every 12 hours if recheck anti-Xa is not at goal) and enoxaparin 30 mg every eight hours; 3) to compare anti-Xa enoxaparin dosing strategies based on VTE, bleeding rates, transfusion requirements, drug discontinuation rate and bioaccumulation, and 4) to determine patient-specific factors that correlate to subtherapeutic anti-Xa such as serial AT-III activity, weight, body mass index, age, cumulative fluid administration, and thromboelastography (TEG).

ELIGIBILITY:
Inclusion Criteria:

* Multi-system trauma
* Anticipated length of stay of at least 72 hours
* At high risk (risk adjustment profile [RAP] >= 5) and initiated on enoxaparin 30 mg every 12 hours per VTE prophylaxis protocol
* No counterindication to trauma team VTE prophylaxis protocol (e.g., intracranial bleeding, incomplete spinal cord injury with hematoma within 24 hours post injury, ongoing hemorrhage, uncorrected coagulopathy, >= grade IV liver or spleen injury, intraocular injury)

Exclusion Criteria:

* Renal dysfunction (creatinine clearance < 30 mL/min or on continuous renal replacement therapy)
* Weight < 50 kg or > 150 kg
* Platelet count < 50,000
* Allergy to heparin or low molecular weight heparin
* On therapeutic anticoagulation on admission or requiring it within 24 hours of admission
* Isolated intracranial hemorrhage
* Known hyperbilirubinemia (serum bilirubin > 6.6 mg/dL)
* Pregnancy
* Incarceration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-03; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Droege, PharmD, Principal Investigator — UC Health - University of Cincinnati Medical Center
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Droege ME, Droege CA, Philpott CD, Webb ML, Ernst NE, Athota K, Wakefield D, Dowd JR, Gomaa D, Robinson BHR, Hanseman D, Elterman J, Mueller EW. Impact of antithrombin III and enoxaparin dosage adjustment on prophylactic anti-Xa concentrations in trauma patients at high risk for venous thromboembolism: a randomized pilot trial. J Thromb Thrombolysis. 2021 Nov;52(4):1117-1128. doi: 10.1007/s11239-021-02478-4. Epub 2021 May 12. PMID 33978907

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1496 screened for eligibility. 1393 excluded.
  51 in control group (anti-Xa 0.1 IU/mL or greater); 52 in intervention group (anti-Xa < 0.1 IU/mL)
  52 patients in the intervention group underwent 1:1 randomization to the two intervention study arms: 26 patients in 40 mg every 12 hours with escalation to 50 mg every 12 hours and 26 patients in 30 mg every 8 hours.
Groups:
- Control Group: Patients with serum anti-Xa level >= 0.1 IU/mL after third dose of enoxaparin 30 mg every 12 hours
  n = 51 4 with AT-III not collected so 47 included in primary outcome analysis
- Intervention Group: Patients with serum anti-Xa < 0.1 IU/mL after third dose of enoxaparin 30 mg every 12 hours
  n = 52
  1 patient withdrew consent; 2 patients did not have AT-III collected. 49 total included in primary outcome analyses.
Period: Primary Endpoint
Arm/Group | Control Group | Intervention Group
Started | 51 | 52
Completed | 47 | 49
Not Completed | 4 | 3
Period: Intervention Group: Randomization
Arm/Group | Control Group | Intervention Group
Started | 0 (Control group patients did not undergo randomization (see study protocol section)) | 52 (52 patients in the intervention group underwent 1:1 randomization to the two intervention study arms: 26 patients in 40 mg every 12 hours with escalation to 50 mg every 12 hours and 26 patients in 30 mg every 8 hours.)
Completed | 0 | 51
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control: Serum Anti-Xa >= 0.1 IU/mL: Patients with serum anti-Xa level >= 0.1 IU/mL after third dose of enoxaparin 30 mg every 12 hours
- Intervention: Serum Anti-Xa < 0.1 IU/mL: Patients with serum anti-Xa level < 0.1 IU/mL after third dose of enoxaparin 30 mg every 12 hours
- Total: Total of all reporting groups
Arm/Group | Control: Serum Anti-Xa >= 0.1 IU/mL | Intervention: Serum Anti-Xa < 0.1 IU/mL | Total
Number analyzed (Participants) | 47 | 51 | 98
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Age | 38 [25 to 58] | 41 [26 to 56] | 41 [26 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 29 | 38 | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Initial AT-III Activity -- Control Group vs. Intervention Group Prior to Randomization
Description: Serum AT-III (% activity) will be compared between the control group and the intervention group patients (combined) after the third dose of enoxaparin 30 mg every 12 hours once initiated at the discretion of the trauma service per current VTE prophylaxis protocol
Time Frame: After third dose of enoxaparin 30mg q12h, which will typically be on Day 2 of enoxaparin
Measure: Median (Inter-Quartile Range); unit: Percent AT-III activity (%)
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 47 | 49
Percent AT-III activity (%) | 87 [80 to 98] | 82 [71 to 96]
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority; p = 0.092, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During patient enrollment up to 28 days, while inpatient
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

LIMITATIONS AND CAVEATS:
Underpowered; See full results and manuscript listed in citation section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT02412982/Prot_SAP_ICF_000.pdf